CLINICAL TRIAL: NCT06529731
Title: A Phase 2 Trial of Interferon-γ (IFN-γ) in Combination With Donor Leukocyte Infusion (DLI) to Treat Relapsed Acute Myeloid Leukemia (AML) and Myelodysplastic Syndromes (MDS) After Allogeneic Hematopoietic Stem Cell Transplantation (alloSCT)
Brief Title: Interferon-γ (IFN-γ) With Donor Leukocyte Infusion to Treat Relapsed Acute Myeloid Leukemia and Myelodysplastic Syndromes Post Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sawa Ito, MD (Other)
Collaborators: Evans MDS Discovery Research Grant (Unknown); Amgen (Industry); FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Sawa Ito, MD, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 23-160; 1R01FD008187-01 (FDA)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: interferon-γ (IFN-γ); donor leukocyte infusion (DLI); allogeneic hematopoietic stem cell transplantation (alloSCT)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IFN-γ + DLI (Experimental): ACTIMMUNE® (IFN-γ-1b) at a dose of 50 mcg/m^2 (All participants will receive a 4-week period of IFN-γ monotherapy with ACTIMMUNE 100 mcg 3 times a week. This dose and schedule will be continued for 4 additional weeks and then tapered to 100 mcg weekly for an additional 4 weeks)
  DLI at a dose of 10^7 CD3+ cells/kg (DLI doses will be given pending clinical assessment for disease, graft versus host disease (GVHD) and peripheral blood donor chimerism the week prior to DLI. Second DLI dose is only offered to subjects with residual disease not requiring cytotoxic therapy and without GVHD)
  Interventions: Drug: Interferon gamma-1b; Biological: Donor Leukocyte Infusion (DLI)

INTERVENTIONS:
Drug: Interferon gamma-1b — ACTIMMUNE/Interferon gamma-1b is a single-chain polypeptide containing 140 amino acids that is produced by fermentation of a genetically engineered Escherichia coli bacterium containing the DNA which encodes for the recombinant protein. Interferon gamma-1b is part of a drug regimen used to treat Chronic Granulomatous Disease, or CGD. CGD is a genetic disorder, usually diagnosed in childhood, that affects some cells of the immune system and the body's ability to fight infections effectively.
  Other Names: ACTIMMUNE®
Biological: Donor Leukocyte Infusion (DLI) — Donor lymphocyte infusion is a procedure that transfers healthy white blood cells (lymphocytes) from a bone marrow or stem cell donor to a recipient's blood. An infusion of healthy lymphocytes helps the recipient's immune system get rid of remaining cancer cells if they have a relapse after a bone marrow or stem cell transplant for blood cancer.

SUMMARY:
This phase 2 study aims to confirm the efficacy seen in the prior phase 1 trial, and further contribute to this effort through the collection of leukemia cells pre- and post- in vivo IFN-γ therapy. As in the previously conducted phase 1 trial, this trial will test whether leukemia blasts were responsive to IFN-γ in vitro and in vivo, with single-cell RNA sequencing (scRNAseq) conducted to understand the transcriptomic changes induced by IFN-γ in leukemia cell subsets, including those with stem cell characteristics.

DETAILED DESCRIPTION:
This novel regimen has the potential to fill a large unmet need for this high-risk population of patients who have few, if any, effective therapeutic options. If this trial confirms the clinical efficacy of IFN-γ/DLI, it will establish a new standard of care for post-transplant AML/MDS relapse. It would also provide a rationale to explore other indications for IFN-γ in the context of an alloSCT, including 1) IFN-γ/DLI for relapsed disease after haploidentical alloSCT; 2) pre-emptive post-alloSCT treatment of patients transplanted with measurable residual disease (MRD) or with poor-risk AML/MDS such as with TP53 mutations; and 3) prevention of relapse in patients who can only tolerate reduced-intensity conditioning regimens which in most studies results in higher rates of post-alloSCT AML/MDS relapse than when intensive conditioning regimens are employed. Together, this work would allow more patients with AML/MDS to be referred for and ultimately benefit from an alloSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Recipients of an alloSCT for AML or MDS from a minimally 8/8 HLA-matched donor
3. AML/MDS relapsed post-alloSCT with measurable residual disease defined by either of the following criteria:

   1. At least 5% or more myeloblasts based on bone marrow biopsy morphology by pathologist review. Abnormal myeloblasts cannot not exceed 30% overall 36
   2. At least 0.1% of abnormal myeloblasts with a leukemia-associated immunophenotype (LAIP) by multiparameter flow cytometry. The abnormal cells with LAIP should not exceed 30% of nucleated cells.
   3. Recurrent or persistent cytogenetic abnormalities detectable by FISH or karyotype analysis.
   4. For patients with mutant NPM1, at least 1,000 mutant transcript copies per 106 ABL or equivalent housekeeping transcripts in bone marrow by qPCR or dPCR
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
5. A DLI is available, or the donor is available and agrees to undergo apheresis to collect lymphocytes for infusion
6. If salvage therapy for post-alloSCT relapse was received, the therapy is limited to 1 line of the following:

   1. For hypomethylating agents, venetoclax, and targeted therapies (e.g., tyrosine kinase inhibitors, IDH1/IDH2 inhibitors, or FLT3 inhibitors), the last dose must be > 2 week prior to the initiation of IFN-γ
   2. For cytotoxic chemotherapy agents, the last dose must be >2 weeks prior to start of treatment for the present study
   3. For investigational agents, the last dose must be ≥ 4 weeks or 5 half-lives (whichever is longer) prior to the start of treatment for the present study
7. Provision of signed and dated informed consent form
8. Stated willingness to comply with all study procedures and availability for the duration of the study
9. For female subject, who is < 55 years old without hysterectomy, oophorectomy or documented menopause, willingness to use two forms of contraception including one form of highly effective contraception (i.e., long-acting reversible contraception, oral contraceptive pills) for the duration of the study
10. For male subject, willingness to use highly effective contraception methods including male condoms by male subject and one form of highly effective contraception by his female partner (i.e., long-acting reversible contraception, oral contraceptive pills) for the duration of the study

Exclusion Criteria:

1. Primary engraftment failure after alloSCT
2. Grade 3 or 4 aGVHD per Mount Sinai Acute GVHD International Consortium (MAGIC) at the time of planned enrollment
3. History of grade 4 aGVHD per the MAGIC criteria
4. Moderate or severe cGVHD per NIH Consensus Criteria at time of planned enrollment
5. Any systemic immunosuppressive medications taken within 2 weeks before the enrollment
6. Grade 3 or higher non-hematologic toxicity related to any prior therapy at the time of enrollment
7. A contraindication to receive IFN-γ including a known hypersensitivity to IFN-γ, E. coli derived products or any other component of the product
8. Positive pregnancy test or currently breastfeeding on Day 1 of study treatment 37
9. Active cardiac arrhythmia not controlled by medical management or current NYHA class II or higher congestive heart failure within 2 months of enrollment unless it was due to a tachyarrhythmia which is under control at the time of enrollment
10. Active ischemic heart disease not controlled with medications within 2 months of enrollment
11. Acute or chronic pulmonary disease requiring continuous oxygen treatment
12. Seizure disorder not controlled by medications within 2 months of enrollment
13. AST or ALT > 5x ULN or total bilirubin >3x ULN at time of enrollment
14. Renal function CrCl <30 mL/min at time of enrollment using modified Cockcroft-Gault formula
15. Body surface area ≤ 1.5 m2 or ≥ 2.5 m2 so as to minimize variation in IFN-γ exposure based on differences in body surface area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | At 1 year
  Occurrence of treatment failure, hematologic relapse from a CR (complete remission)/CRh/Cri), or death observed from start of IFN-γ treatment. Patients alive at 1 year after start of treatment will be censored on the date of last contact.

SECONDARY OUTCOMES:
Event-free survival (EFS) - Landmark 1-year | Up to 1 year
  Time from start of IFN-γ treatment until event of death, date of treatment failure, or hematologic relapse from a CR/CRh/Cri. CR is defined by blasts less than 5% by morphology defined by bone marrow blasts less than 5%; absence of circulating blasts; absence of extramedullary disease; absolute neutrophil count (ANC) at or greater than 1,000/mL; platelet count at or greater than 100,000/mL CRh is defined by ANC at or greater than 500/mL and platelet count at or greater than 50,000/mL otherwise all other CR criteria met. CRi is defined by all CR criteria except for residual neutropenia less than 1,000/mL or thrombocytopenia less than 100,000/mL Treatment failure is not achieving either CR, CRh or CRi by 6 months. Patients evaluable for response without CR, CRh or CRi by 6 months and patients who die before 6 months without response assessments are considered an event at day 1 of IFN-γ treatment
Minimal residual disease (MRD) | At 6 months
  Rate of complete remission (CR) with no measurable disease at 6 months. CR is defined as
Complete Remission (CR) | At 6 months
  Proportion of patients who experience Complete Remission (CR). CR is defined by bone marrow blasts less than 5%; absence of circulating blasts; absence of extramedullary disease; absolute neutrophil count (ANC) at or greater than 1,000/mL; platelet count at or greater than 100,000/mL. The proportion of responders will be calculated as the number of responders divided by the number of evaluable patients.
Complete remission with partial hematologic recovery (CRh) | At 6 months
  Proportion of patients who experience Complete remission with partial hematologic recovery (CRh). CRh is defined by ANC at or greater than 500/mL and platelet count at or greater than 50,000/mL otherwise all other CR criteria met. The proportion of responders will be calculated as the number of responders divided by the number of evaluable patients.
Complete remission with incomplete count recovery (CRi) | At 6 months
  Proportion of patients who experience complete remission with incomplete count recovery (CRi). CRi is defined by all CR criteria except for residual neutropenia less than 1,000/mL or thrombocytopenia less than 100,000/mL51. The proportion of responders (CR, CRh, or CRi) will be calculated as the number of responders divided by the number of evaluable patients. The proportion of responders will be calculated as the number of responders divided by the number of evaluable patients.
Overall survival | Up to 1 year
  Time from start of IFN-γ to death by any cause or censored on the date of last contact.
Rate of donor chimerism | At 6 months
  Proportion of the efficacy population with ≥95% peripheral blood CD3+ and CD33+ cells and of unfractionated bone marrow being donor-derived
Rate of transfusion independence | At 1 year
  Proportion of the subjects who achieve the absence of a red-cell or platelet transfusion for at least 56 days between the first and last day of treatment.
Frequency and severity of adverse events (AEs) | Up to 6 months
  Number of patients who experience an Adverse Event or Serious Adverse Event related to study treatment, per CTCAE v5.0 criteria. Distinct number of patients will be determined per each event type by highest grade experienced.
Frequency of new onset grade 3 or 4 acute graft-versus-host disease (aGVHD) | Up to 12 months
  number of patients meeting criteria for grade 3 or 4 aGVHD per MAGIC divided by the number of evaluable patients. The MAGIC criteria as follows: Overall clinical grade (based on most severe target organ involvement): Grade 0: No stage 1-4 of any organ; Grade I: Stage 1-2 skin without liver, upper GI, or lower GI involvement; Grade II: Stage 3 rash and/or stage 1 liver and/or stage 1 upper GI and/or stage 1 lower GI; Grade Ill: Stage 2-3 liver and/or stage 2-3 lower GI, with stage 0-3 skin and/or stage 0-1 upper GI; Grade IV: Stage 4 skin, liver, or lower GI involvement, with stage 0-1 upper GI.
Frequency of new onset moderate or severe chronic GVDH (cGVHD) | Up to 12 months
  The number of patients meeting criteria for moderate or severe cGVHD per NIH Consensus Criteria divided by the number of evaluable patients. The NIH Consensus Criteria is a diagnostic assessment that evaluates hair, skin, nails, eyes, mouth, genitalia, GI tract, liver, lung, muscles and joints, hematopoietic and immune system, cardiac and neurological condition/function, to determine whether or not the GVHD is chronic.

CONTACTS AND LOCATIONS:
Overall Officials: Sawa M Ito, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (3):
- United States (3):
  - Washington University, St Louis, Missouri
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No